CLINICAL TRIAL: NCT02626416
Title: Self-monitoring of Visual Axis Opacification (VAO) Under Non-clinical Settings in China
Brief Title: Monitoring of Visual Axis Opacification Under Non-clinical Settings
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Haotian Lin, Principal Investigator, Home for Cataract Children, Zhongshan Ophthalmic Center, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CCPMOH2010-China10
Record Dates: First submitted 2015-12-07; First posted 2015-12-10 (Estimated); Last update posted 2015-12-10 (Estimated); Status verified 2015-12

CONDITIONS: Cataract
Keywords: Telemedicine
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- telemedicine group (Experimental): Congenital cataract patients use telemedicine to pursue and adjust the time of follow-up under non-clinical settings
  Interventions: Device: LenZOC (mobile application)
- non-telemedicine group (No Intervention): Congenital cataract patients pursue and adjust the time of follow-up through outpatient visit in the hospital

INTERVENTIONS:
Device: LenZOC (mobile application) — The transparency of the visual axial at the anterior segment is observed through a dilated pupil. Image of the eye of a patient taken with LenZOC is calibrated with a standardized white and black bar adhered to the patient's eyelid. Calibrated images are dimmed as graysalegrayscale. The intensity and progress of visual axial opacification (VAO) is quantified as absolute area and relative area (calculated as: absolute area of VAO/ absolute area of dilated pupil).
  Arms: telemedicine group

SUMMARY:
The incidence rate of postoperative capsular opacification (PCO) in children after cataract surgery is reported to be as high as 100%, while timely Nd: YAG laser posterior capsulotomy is effective to treat visual axis opacification (VAO) caused by PCO. Therefore, long-term follow-up, timely diagnosis and treatment is important to improve patient's outcome.

The major and central part of lens is easy to be observed through a dilated pupil. Especially, opacification in the lens and/or lens capsule is distinctive showing as "white" on the "black" background. The characteristic features of the disease and advances in photographic technique with mobile phone make it possible for patients and/or their guardians to monitor the progress of cataract or PCO with mobile application in a "self-help" manner under non-clinical settings.

DETAILED DESCRIPTION:
The incidence rate of postoperative capsular opacification (PCO) in children after cataract surgery is reported to be as high as 100%, while timely Nd: YAG laser posterior capsulotomy is effective to treat visual axis opacification (VAO) caused by PCO. Therefore, long-term follow-up, timely diagnosis and treatment is important to improve patient's outcome.

The major and central part of lens is easy to be observed through a dilated pupil. Especially, opacification in the lens and/or lens capsule is distinctive showing as "white" on the "black" background. The characteristic features of the disease and advances in photographic technique with mobile phone make it possible for patients and/or their guardians to monitor the progress of cataract or PCO with mobile application in a "self-help" manner under non-clinical settings. In this way, patients and/or guardians could adjust the time of return to clinical follow-up visit accordingly. Furthermore, standardized and analyzed pictures could be sent to clinicians for remote diagnosis when necessary.

The investigators developed a mobile phone application LenZOC. The investigators aimed to assess whether mobile phone application for parents of children with cataracts would improve their adherence with follow-up and increase rates of timely detection and management of treatable conditions such as posterior capsular opacification (PCO).

ELIGIBILITY:
Inclusion Criteria:

* Children after cataract surgery for more than 1 year without any postoperative complications
* Without other ocular abnormality
* Parents owned a smart mobile phone that meets the requirements for installation of the LenZOC
* Written informed consents provided

Exclusion Criteria:

* Intraocular pressure >21 mmHg
* Pre-existing ocular diseases including but not restricted to:

Glucoma Micro-cornea Micro-ophthalmic Diseases of post-segment that might lead to VAO

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 1400 (Estimated)
Dates: Start 2016-01; Primary Completion 2018-01 (Estimated); Study Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
Times of follow-ups for each participant | up to one year

SECONDARY OUTCOMES:
Best corrected visual acuity | up to 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Haotian Lin, M.D. Ph.D., Principal Investigator — Zhongshan Ophthalmic Center, Sun Yat-sen University; Yizhi Liu, M.D. Ph.D., Study Chair — Zhongshan Ophthalmic Center, Sun Yat-sen University; Weirong Chen, M.D., Study Director — Zhongshan Ophthalmic Center, Sun Yat-sen University
Locations (1):
- Zhognshan Ophthalmic Center, Sun Yat-sen University, Guangzhou, Guangdong, China

REFERENCES:
- [Background] Lin H, Chen W, Luo L, Congdon N, Zhang X, Zhong X, Liu Z, Chen W, Wu C, Zheng D, Deng D, Ye S, Lin Z, Zou X, Liu Y. Effectiveness of a short message reminder in increasing compliance with pediatric cataract treatment: a randomized trial. Ophthalmology. 2012 Dec;119(12):2463-70. doi: 10.1016/j.ophtha.2012.06.046. Epub 2012 Aug 24. PMID 22921386
- [Background] Rivas-Perea P, Baker E, Hamerly G, Shaw BF. Detection of leukocoria using a soft fusion of expert classifiers under non-clinical settings. BMC Ophthalmol. 2014 Sep 9;14:110. doi: 10.1186/1471-2415-14-110. PMID 25204762
- [Background] Lin H, Long E, Chen W, Liu Y. Documenting rare disease data in China. Science. 2015 Sep 4;349(6252):1064. doi: 10.1126/science.349.6252.1064-b. No abstract available. PMID 26339020
- [Background] Plager DA, Lynn MJ, Buckley EG, Wilson ME, Lambert SR; Infant Aphakia Treatment Study Group. Complications, adverse events, and additional intraocular surgery 1 year after cataract surgery in the infant Aphakia Treatment Study. Ophthalmology. 2011 Dec;118(12):2330-4. doi: 10.1016/j.ophtha.2011.06.017. Epub 2011 Sep 16. PMID 21925737
- [Background] Rong X, Ji Y, Fang Y, Jiang Y, Lu Y. Long-Term Visual Outcomes of Secondary Intraocular Lens Implantation in Children with Congenital Cataracts. PLoS One. 2015 Jul 31;10(7):e0134864. doi: 10.1371/journal.pone.0134864. eCollection 2015. PMID 26230501
- See also: Home Page of Zhongshan Ophthalmic center — http://www.gzzoc.com